CLINICAL TRIAL: NCT05879354
Title: Investigation of the Effect of Active Cycle of Breathing Techniques on Respiratory Distress Symptom Cluster in Patients With Lung Cancer
Brief Title: Active Cycle of Breathing Techniques on Respiratory Distress Symptom Cluster
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Doğa Ulcay, Lecturer, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MAU_DogaUlcay_001
Record Dates: First submitted 2023-04-13; First posted 2023-05-30 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Lung Neoplasms
Keywords: Active Cycle of Breathing Techniques; Lung Neoplasms; Symptom Cluster; Nursing; Care
MeSH Terms: conditions — Lung Neoplasms; Syndrome

STUDY DESIGN:
Intervention Model Description: The intervention group will apply the Active Cycle of Breathing Techniques with video twice a day for 28 days and the control group will not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Cycle Of Breathing Techniques Group (Experimental): Patients in the intervention group will be provided with video-guided Active Cycle of Breathing Techniques twice a day for 28 days.
  Interventions: Other: Active Cycle of Breathing Techniques
- Control group (No Intervention): No intervention will be given to the patients in the control group.

INTERVENTIONS:
Other: Active Cycle of Breathing Techniques — Patients in the intervention group will be provided with video-guided Active Cycle of Breathing Techniques twice a day for 28 days.
  Arms: Active Cycle Of Breathing Techniques Group

SUMMARY:
This study was designed as a randomized, control group, experimental study to examine the effect of Active Cycle of Breathing Techniques application on respiratory distress symptom cluster in patients with lung cancer.

DETAILED DESCRIPTION:
The sample of the study will consist of patients who received chemotherapy treatment with the diagnosis of Stage IV non-small cell lung cancer in the outpatient chemotherapy service of a training and research hospital and met the inclusion criteria. Data in the study will be collected using the Patient Information Form, Eastern Cooperative Oncology Group (ECOG) Performance Scale, Cancer Dyspnea Scale, Leicester Cough Questionnaire and Cancer Fatigue Scale. In order to test the applicability and comprehensibility of the forms to be used before the study, a preliminary application will be made with 5 patients. This study is planned to prepare a video describing the application for patients to use while performing the Active Cycle of Breathing Techniques application. On the 1st day of the study, a 10-minute face-to-face training will be given to the intervention (experimental) group by the researcher using the video about the Active Cycle of Breathing Techniques. In the research, the intervention (experimental) group will be asked to follow the video to be prepared and apply the Active Cycle of Breathing Techniques twice a day for 28 days. The intervention (experimental) group will be monitored by telephone call once a week and 3 times using the Patient Follow-up Form (days 7, 14 and 21). On the other hand, only the pre-test and post-test will be applied to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Being diagnosed with stage IV non-small cell lung cancer
* Being diagnosed with lung cancer in the type of adenocarcinoma and squamous cell carcinoma
* Receiving outpatient chemotherapy treatment
* Receiving the first course of chemotherapy treatment
* ECOG Performance Scale Score < 3
* Having all the symptoms of dyspnea, cough, and fatigue
* Not having a cognitive disorder or a diagnosed psychiatric illness
* Being able to speak Turkish
* Volunteering to participate in the research

Exclusion Criteria:

* Experiencing a chronic obstructive pulmonary disease (COPD) exacerbation in the last 4 weeks
* Having an active lung infection
* Not volunteering to participate in the research
* Not having dyspnea, cough, and fatigue symptoms
* Not speaking Turkish

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Dyspnea Level | 28 Days
  The level of dyspnea will be lower in patients in the intervention (experimental) group to whom Active Breathing Cycle techniques were applied, compared to the patients in the control group who did not. The Turkish version of the Cancer Dyspnea Scale, the Turkish Validity and Reliability of which was made by Bitek and Tokem in 2021, will be used to measure the level of dyspnea.
Fatigue Level | 28 days
  The level of fatigue will be lower in patients in the intervention (experimental) group to whom Active Breathing Cycle techniques were applied, compared to the patients in the control group who did not. The Turkish version of the Hirai Cancer Fatigue Scale, the Turkish validity and reliability of which was made by Mencel in 2021, will be used to measure the level of fatigue.
Health-related quality of life in chronic cough | 28 days
  The level of health-related quality of life in chronic cough will be lower in patients in the intervention (experimental) group to whom Active Breathing Cycle techniques were applied, compared to the patients in the control group who did not. The Turkish version of the Leicester Cough Questionnaire (LCQ), the Turkish validity and reliability of which was made by Gonen ve Havlucu in 2014, will be used to measure the level of health-related quality of life in chronic cough.

CONTACTS AND LOCATIONS:
Overall Officials: Doğa Ulcay, Msc, Principal Investigator — Maltepe University; Semiha Akın, Prof., Principal Investigator — University of Health science; Akın Öztürk, Specialist, Principal Investigator — Süreyyapaşa Chest Diseases and Thoracic Surgery Training And Research Hospital
Locations (1):
- Süreyyapaşa Chest Diseases and Thoracic Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)